CLINICAL TRIAL: NCT03581565
Title: Effect of Cementation Technique Applied for Single-tooth Implant Crowns on Residual Cement: A Three-arm Parallel-group Randomized Clinical Trial
Brief Title: Cementation Techniques for Single-tooth Implant Crowns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kıvanç Akça (Other)
Collaborators: Hacettepe University (Other)
Responsible Party: Sponsor-Investigator, Kıvanç Akça, Prof. Dr., Hacettepe University
Organization: Hacettepe University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: KA-17043; THD-2018-16143 (Other Grant/Funding Number: HacettepeU Scientific Research Projects Coordination Unit)
Record Dates: First submitted 2018-06-06; First posted 2018-07-10 (Actual); Last update posted 2018-07-10 (Actual); Status verified 2018-06

CONDITIONS: Cementation (MeSH Unique ID: D002484); Dental Implant-Abutment Design (MeSH Unique ID: D059605); Crown (MeSH Unique ID: D003442) Surfaces; Contour: Crown (MeSH Unique ID: D003442) - Dental Implant (MeSH Unique ID: D015921) Abutment
Keywords: cementation; dental implant; crown; periimplantitis
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Technique I (Active Comparator): Loading of a zinc polycarboxylate (with the requirements of ISO 9917) cement to fulfill the crown
  Cement: Poly-F, DentsplySirona, York, Pennsylvania, United States Mixing Ratio: 1 scoop powder: 2 drops liquid Mixing Time (extraoral): 30 seconds Working Time (extraoral): 45 seconds Application (extraoral): placement of mixture into crown using a heidemann Spatula Setting Time (intraoral): 2-8 minutes
  Interventions: Other: zinc polycarboxylate (with the requirements of ISO 9917)
- Technique II (Active Comparator): Loading of a zinc polycarboxylate (with the requirements of ISO 9917) to fill the coronal half of the crown
  Cement: Poly-F, DentsplySirona, York, Pennsylvania, United States Mixing Ratio: 1 scoop powder: 2 drops liquid Mixing Time (extraoral): 30 seconds Working Time (extraoral): 45 seconds Application (extraoral): placement of mixture into crown using a heidemann Spatula Setting Time (intraoral): 2-8 minutes
  Interventions: Other: zinc polycarboxylate (with the requirements of ISO 9917)
- Technique III (Active Comparator): Application of a zinc polycarboxylate (with the requirements of ISO 9917) to the axial walls of internal surface of crown
  Cement: Poly-F, DentsplySirona, York, Pennsylvania, United States Mixing Ratio: 1 scoop powder: 2 drops liquid Mixing Time (extraoral): 30 seconds Working Time (extraoral): 45 seconds Application (extraoral): application of mixture into crown using a bonding applicator tip Setting Time (intraoral): 2-8 minutes
  Interventions: Other: zinc polycarboxylate (with the requirements of ISO 9917)

INTERVENTIONS:
Other: zinc polycarboxylate (with the requirements of ISO 9917) — intraoral cementation of single-tooth implant crowns with three different technique, intraoral removal of cement excess upon setting

SUMMARY:
Cement retention has been widely used for implant-supported fixed partial dentures in daily dental practice. The cementation approach indeed offers straightforward clinical application protocol which is basically conceptualized for tooth/teeth supported fixed restorations. However, removal of excess cement around implant restorations presents specific difficulties. More importantly, there are certain biological consequences due to residual cement leftover in peri-implant sulcus. There is no evidence based guidance with regards to cementation techniques applied for implant supported fixed restorations due to limited clinical studies. Therefore the aim of this clinical trial is to compare three different cementation technique with regards to removal of excess cement and other clinical subsidiaries (abutment margin, crown surface and contour) involving indirectly as well.

DETAILED DESCRIPTION:
Single-tooth implant crowns to replace missing molar tooth were addressed to qualify and quantify residual cement on implant-abutment complex and peri-implant soft tissue following cementation. Thirty bone-level dental implants of one kind enrolled in the study. Prior to delivery of screw-retained crowns completed for usual treatment, implants were allocated randomly to a trial comparison group. Three different cement loading approach, ten in each group, was applied using cement-retained trial crowns on prefabricated metal abutments. Following completion of the assigned cementation technique, the trial crown was removed with its abutment accessing from the occlusal hole prepared after removal of excess cement. Then, the presence of residual cement on implant-abutment complex and implant soft tissue in accordance with axial and proximal surfaces was qualified. To quantify the amount of residual cement in accordance with location and distribution, the crown-abutment complex was digitized three-dimensionally using an intra-oral scanner. The output of surface data was evaluated in virtual 3-D image for cement excess, when detected location in the abutment-crown complex is recorded, area and distribution was calculated using a software. The frequency of occurrence and quantity of residual cement of 3-different cementation techniques was statistically evaluated using logistic and linear regression model separately considering abutment margin, crown surface and contour.

ELIGIBILITY:
Inclusion Criteria:

* completed growth and development
* periodontally and dentally healthy conditions
* missing single molar tooth without free-end edentulism
* bone-level standard diameter of a specific implant from one manufacturer
* complication free healing period for osseointegration following straightforward surgical implant placement
* natural dentition or fixed restoration in dental arch
* signing of informed consent form

Exclusion Criteria:

* absolute systemic contraindications for implant surgery (e.g. bone cancer, radiation therapy)
* relative systemic contraindications for implant surgery (e.g. diabetes, steroid therapy)
* risk factors (e.g. smoking, limited mouth opening)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-10-16 (Actual); Primary Completion 2018-03-19 (Actual); Study Completion 2018-05-25 (Actual)

PRIMARY OUTCOMES:
visual assessment of residual cement on crown-abutment complex | 15 minutes
  removal of cemented crown-abutment complex to detect excess cement on the mesial, distal, buccal and lingual surfaces of crown and abutment separately scoring: presence or absence
measurement of residual cement area and distribution | 30 minutes
  digitalization of the removed crown-abutment complexes those scored with cement presence, then using a software, virtual selection of existing cement to calculate the area in millimeter square and to define the direction and the extension in millimeters on the mesial, distal, buccal and lingual surfaces of crown and abutment separately

SECONDARY OUTCOMES:
visual assessment of residual cement around the peri-implant soft tissue | 15 minutes
  removal of cemented crown-abutment complex to detect excess cement on the peri-implant soft tissue contacting the mesial, distal, buccal and lingual surfaces of crown-implant complex scoring: presence or absence

OTHER OUTCOMES:
correlation of abutment margin and crown-abutment contour with 'Outcome 2' measures | 30 minutes
  Recording of stock abutment margin location at mesial, distal, buccal and lingual surfaces in relation to peri-implant soft tissue level measurement in millimeters
  Defining of abutment to crown transition angle at mesial, distal, buccal and lingual surfaces description as concave, convex or flat
recognition of residual cement on radiographs | 20 minutes
  evaluation of peri-apical radiographs of cemented crowns to detect presence of excess cement on mesial and distal surfaces scoring: presence or absence

CONTACTS AND LOCATIONS:
Overall Officials: Kıvanç Akça, Prof.Dr., Study Director — Hacettepe University
Locations (1):
- Hacettepe University Faculty of Dentistry Department of Prosthodontics, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No